CLINICAL TRIAL: NCT02164110
Title: A Randomized, Single Blind, Multicenter, Therapeutic Confirmatory Study to Assess the Efficacy (Immunogenicity) and Safety of Euvichol in Healthy Adults and Children
Brief Title: To Evaluate the Efficacy (Immunogenicity) and Safety of Euvichol in Healthy Adults and Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EuBiologics Co.,Ltd (Industry)
Collaborators: Instituto Universitario IVI (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UBC301
Record Dates: First submitted 2014-04-27; First posted 2014-06-16 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Prevention Harmful Effects
MeSH Terms: interventions — shanchol; Cholera Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Euvichol (Experimental): * Number of doses and intervals: two doses/Weeks 0 and 2
  * Method of administration: oral administration
  * Dose of drug to be administered: 1.5 mL/dose
  Interventions: Biological: Euvichol
- Shanchol (Active Comparator): * Number of doses and intervals: two doses/Weeks 0 and 2
  * Method of administration: oral administration
  * Dose of drug to be administered: 1.5 mL/dose
  Interventions: Biological: Shanchol

INTERVENTIONS:
Biological: Euvichol — * Number of doses and intervals: two doses/Weeks 0 and 2
  * Method of administration: oral administration
  * Dose of drug to be administered: 1.5 mL/dose
  Other Names: Oral Cholerae Vaccine
  Arms: Euvichol
Biological: Shanchol — * Number of doses and intervals: two doses/Weeks 0 and 2
  * Method of administration: oral administration
  * Dose of drug to be administered: 1.5 mL/dose
  Other Names: Oral cholera vaccine
  Arms: Shanchol

SUMMARY:
The purpose of this study is to evaluate the efficacy (Immunogenicity) and Safety of Euvichol in Healthy Adults and Children.

DETAILED DESCRIPTION:
A randomized, single blind, multicenter, therapeutic confirmatory study to assess the efficacy (immunogenicity) and safety of Euvichol in healthy adults and children

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to study participation voluntarily provided by an individual or his/her legally acceptable representative.
2. Age of 1 ~ 40 years
3. An individual who can be followed up during the study period and is capable of complying with the study requirements.

Exclusion Criteria:

1. History of hypersensitivity reactions to other preventative vaccinations.
2. Immune function disorders including immunodeficiency diseases.
3. An individual thought to have difficulty participating in the study due to severe chronic diseases, based on the judgment of the investigator.
4. 38℃ or higher body temperature measured prior to investigational product dosing.
5. Abdominal pain, nausea, vomiting, or decreased appetite within 24 hours prior to study initiation.
6. Diarrhea or administration of antidiarrheal drugs or antibiotics to treat diarrhea within 1 week prior to study initiation.
7. Other vaccination within 1 week prior to study initiation or planned vaccination during the study.
8. Diarrhea or abdominal pain lasting 2 weeks or longer within 6 months prior to study initiation.
9. Participation in another clinical trial with investigational product dosing within 1 month prior to study initiation.
10. Pregnant or lactating women.
11. An individual thought to have difficulty participating in the study due to other reasons, based on the judgment of the investigator
12. Applicable to the Pivotal study only: history of cholera vaccinations or history of cholera.

Ages: 1 Year to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3632 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Efficacy | 14 days after second doses
  Proportion of subjects exhibiting 4-fold or greater rises in titers of anti-V. cholera O1 antibody, relative to baseline
Safety | From first shot to 14 days after second dose
  Type and frequency of solicited adverse event type (Day 0 ~ 6), Type and frequency of unsolicited adverse event type (Day 0 ~ Day 28)

SECONDARY OUTCOMES:
Efficacy | 14 days after second doses
  1. Proportion of subjects exhibiting 4-fold or greater rises in titers of anti-V. cholera O139 antibody, relative to baseline
Safety | From first shot to 14 days after second dose
  1. Change from baseline in vital signs and physical examination
Efficacy | 14 days after second doses
  1. Geometric Mean Titer (GMT) and Geometric Mean Ratio (GMR) as measured by each anti-V. cholera antibody titer at Week 2 (Visit 3) after the second dose as compared to prior to investigational product dosing (Visit 1).
Safety | 14 days after second doses
  1. Change from baseline in laboratory tests (hematologic test, blood chemistry test, urinalysis) to be performed only in subjects who participate in the Pivotal study.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto A. Espos, MD, Principal Investigator — De La Salle University Hospital Medical Center
Locations (1):
- Antonio D. Ligsay, MD, Quezon City, Philippines